CLINICAL TRIAL: NCT03583736
Title: Rapid First Contact Using Virtual Visits to Improve Time-To-Treatment for Patients With Uterine Cancer
Brief Title: Rapid First Contact Using Virtual Visits to Improve Time-To-Treatment for Uterine Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decision
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3818
Record Dates: First submitted 2018-06-27; First posted 2018-07-11 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — Office Visits

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid first contact virtual visit (Active Comparator): Subjects will accept the offer of a virtual visit after being contacted by the nurse to offer a virtual visit with the oncologist prior to the in person office visit once a diagnosis has been confirmed. Subjects will be randomized after accepting offer of a virtual visit.
  Interventions: Behavioral: Virtual visit
- First contact in person office visit (Placebo Comparator): Subjects will accept the offer of a virtual visit after being contacted by the nurse to offer a virtual visit with the oncologist prior to the in person office visit once a diagnosis has been confirmed. Subjects will be randomized after accepting offer of a virtual visit.
  Interventions: Behavioral: Office visit

INTERVENTIONS:
Behavioral: Virtual visit — Virtual visit with oncologist following uterine cancer diagnosis prior to scheduled office visit.
  Arms: Rapid first contact virtual visit
Behavioral: Office visit — Scheduled office visit with oncologist following uterine cancer diagnosis.
  Arms: First contact in person office visit

SUMMARY:
This project aims to evaluate whether rapid first contact with the oncologist the same day or the next day after pathologic diagnosis contributes to a decreased time to treatment, decreased patient anxiety and increased patient satisfaction.

DETAILED DESCRIPTION:
Time to treatment (time from disease diagnosis to initiation of treatment) impacts outcomes in uterine cancer. When controlled for stage, patients with longer time to treatment tend to have less favorable outcomes. Similarly, longer time to treatment has a negative impact on patients' quality of life and markers for anxiety. Our experience at this institution suggests that the time to referral (time from uterine cancer diagnosis and the patients' first encounter with the oncologist) is variable and presents the greatest opportunity for decreasing time to treatment. Among the factors that contribute to the time to referral are the time taken by the referring provider to relay the diagnosis to the patient, time taken to schedule an appointment with the specialist, and the patient's availability to keep an appointment.

Virtual visits provide an opportunity to expedite consultation with the treating oncologist by removing some of the barriers that delay face-to-face visits. Among these barriers are patients' availability for a short notice face-to-face visit based on their work or family obligations, access to transportation, and mental preparedness.

ELIGIBILITY:
Inclusion Criteria:

* Uterine cancer diagnosis on biopsy read by Cleveland Clinic Pathology Department
* Patients must be willing to participate in a virtual visit as the initial meeting with an oncologist at the Cleveland Clinic.
* Receive care at Fairview Hospital, Hillcrest Hospital or Cleveland Clinic Main Campus
* Internet connected smartphone or internet connected computer with webcam
* Participants must have email access
* English speaking
* Competent to make clinic decisions

Exclusion Criteria:

* No diagnosis of uterine cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to treatment following diagnosis to treatment initiation | 30 days
  How long between diagnosis to treatment

SECONDARY OUTCOMES:
Amount of anxiety demonstrated when virtual visits are added | 30 days
  Level of anxiety using GAD-7
Number of patients willing to pay for a virtual visit | 30 days
  Assess patients valuation of virtual visits by measuring their willingness to pay
Number of patients with improved satisfaction scores | 30 days
  Determine whether the addition of a rapid virtual visit improves patients satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jason Knight, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center